CLINICAL TRIAL: NCT03530930
Title: Analgesic, Antiinflammatory and Metabolic Effects of Comarum Palustre in Patients With Osteoarthritis and Diabetes Mellitus
Brief Title: Comarum Palustre in Knee Osteoarthritis and Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal State Budgetary Scientific Institution, Research Institute of Fundamental and Clinical Immunology (Other)
Responsible Party: Principal Investigator, Ivan Shirinsky, MD, PhD, Principal Investigator, Federal State Budgetary Scientific Institution, Research Institute of Fundamental and Clinical Immunology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCI001
Record Dates: First submitted 2017-12-07; First posted 2018-05-21 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Osteoarthritis; Diabetes Mellitus
MeSH Terms: conditions — Osteoarthritis; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comarum Palustre (Experimental): Patients taking Comarum Palustre together with conventional treatment for osteoarthritis
  Interventions: Drug: Comarum Palustre

INTERVENTIONS:
Drug: Comarum Palustre — Comarum Palustre tablets 500 mg BID, 1 month
  Other Names: Potentilla palustris

SUMMARY:
The study evaluates analgesic, antiinflammatory and metabolic effects of Comarum palustre in patients with knee osteoarthritis (OA) and diabetes mellitus. Patients with osteoarthritis will receive Comarum palustre together with conventional treatment of osteoarthritis and diabetes.

DETAILED DESCRIPTION:
Comarum palustre have been shown to exert analgesic properties in patients with knee osteoarthritis not responding to diclofenac. In animal models comarum palustre showed anti-inflammatory, immunomodulatory, analgesic, antioxidant, antihistamine, and membrane-stabilizing effects. Thus, pleiotropic properties of Comarum Palustre may provide a rationale for this use in patients having both osteoarthritis and diabetes mellitus. In this group of patients Comarum Palustre may not only relieve OA-related pain but reduce systemic inflammation, decrease progression of atherosclerosis and diabetes complications.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of the knee fulfilling American College of Rheumatology (ACR) criteria
* diagnosis of type 2 diabetes mellitus

Exclusion Criteria:

* use of NSAIDs one month prior to study entry (paracetamol is allowed)
* pregnancy and lactation
* increased sensitivity to the study drug
* clinically significant renal function impairment
* use of antidepressants
* diagnosis of bipolar disorder
* use of symptomatic slow acting drugs of OA (SYSADOA) one month prior to study entry
* any condition which may lead to difficulties to participation in the study from the viewpoint of Investigator

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2018-11-25 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Visual Analogue Scale for Pain | Baseline, 4 weeks
  The Visual Analogue Scale for Pain varies from 0 to 10 cm. Higher values represent worse outcomes.

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) - subscale Pain | Baseline, 4 weeks
  KOOS Pain consists of 9 items, which are answered on a 4-point likert scale (0=no problems, 4=extreme problems). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Knee injury and Osteoarthritis Outcome Score (KOOS) - subscale Activities of daily living (ADL) | Baseline, 4 weeks
  KOOS ADL consists of 17 items, which are answered on a 4-point likert scale (0=no problems, 4=extreme problems). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Knee injury and Osteoarthritis Outcome Score (KOOS) - subscale Symptoms | Baseline, 4 weeks
  KOOS Symptoms consists of 7 items, which are answered on a 4-point likert scale (0=no problems, 4=extreme problems). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Quality of life with the The Short Form (36) Health Survey score | Baseline, 4 weeks
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section.Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Intermittent and Constant Osteoarthritis Pain self-report questionnaire | Baseline, 4 weeks
  Pain measure: Scale range 0-100 with higher scores indicating worse pain
Changes in serum levels of aggrecan | Baseline, 4 weeks
  serum levels of aggrecan measured in ng/ml
Changes in serum levels of antibodies to collagen type II | Baseline, 4 weeks
  serum levels of antibodies to collagen type II measured AU/ml
Changes in serum levels of C-reactive protein | Baseline, 4 weeks
  serum levels of C-reactive protein (CRP), g/l
Changes in histamine levels | Baseline, 4 weeks
  serum levels of histamine in ng/ml
Changes in inflammation biomarkers | Baseline, 4 weeks
  serum levels of (CRP), interleukin (IL)-6, IL- 18, adiponectin, IL-10, and interferon (IFN) γ in pg/ml
Changes in neopterin levels | Baseline, 4 weeks
  serum neopterin measured in nmol/L
Changes in lipid biomarkers | Baseline, 4 weeks
  serum total cholesterol, HDL, and LDL measured in mmol/L
changes in diabetes control | Baseline, 4 weeks
  Glycated haemoglobin (HbA1c)
Changes in depression scores measured with Patient Health Questionnaire-9 (PHQ9P) | Baseline, 4 weeks
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. It consists of nine questions with responses ranging from "0" (not at all) to "3" (nearly every day). The possible range is 0-27. Higher values represent worse outcome.
Patient global assessment of osteoarthritis | Baseline, 4 weeks
  The Visual Analogue Scale for the Patient global assessment of osteoarthritis varies from 0 to 10 cm. Higher values represent worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Shirinsky, Principal Investigator — Federal State Budgetary Scientific Institution, Research Institute of Fundamental and Clinical Immunology
Locations (1):
- Laboratory of Clinical Immunopharmacology, Novosibirsk, Russia